CLINICAL TRIAL: NCT03469128
Title: Cognitive Processing Therapy Versus Sertraline for the Treatment of Post-traumatic Stress Disorder & Substance Use Disorder Egyptian Patients
Brief Title: Cognitive Processing Therapy vs. Sertraline for the Treatment of PTSD & SUD in Egyptian Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Amani Safwat Albrazi, Principal Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2016-2017PTBUE; IRB Protocol CL-006 (Registry Identifier: the British University in Egypt Institutional Review Board)
Record Dates: First submitted 2018-01-31; First posted 2018-03-19 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Psychologic Manipulation
Keywords: PTSD; CPT; SUD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sertraline

STUDY DESIGN:
Intervention Model Description: Data were obtained by interviewing 587 patients diagnosed with SUD. Patients were interviewed by a clinician and asked to complete: Mini-International Neuropsychiatric Interview (M.I.N.I), and Clinician-Administered PTSD Scale (CAPS). Patients with comorbid SUD and PTSD were asked to complete: The Brief Addiction Monitor (BAM), PTSD Checklist-Civilian (PCL-5), Beck Depression Inventory (BDI-II), and Timeline Follow Back Interview (TLFB). Patients with comorbid SUD and PTSD were randomized to one of the following groups: 1) received CPT. 2) received Sertraline. 3) the Placebo control group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This is a three-group, repeated-measure, parallel-group, Randomized Control Trial design. Patients, study psychiatrists, and assessors were blind to treatment condition assignment. Randomization blocks of three were used to maintain equal group size. The 3-month assessment serves as the post-treatment. Outcome assessments were PTSD severity, substance use severity, and depression. The pharmacy of Ain Shams Hospital created sertraline and matching placebo kits with single-identifier numbers based on a random code that was provided to an unblinded statistician who will instruct the psychiatrist how to distribute kits to patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive processing therapy (Active Comparator): Cognitive Processing Therapy (CPT) in which participants completed 12 sessions of CPT
  Interventions: Behavioral: Cognitive processing therapy
- Sertraline (Active Comparator): Patients with co-occurrence PTSD & SUD disorders were treated by Sertraline.
  Interventions: Drug: Sertraline
- Control group (Placebo Comparator): Placebo Control group
  Interventions: Other: Placebo Control

INTERVENTIONS:
Behavioral: Cognitive processing therapy — Psychological treatment for patients suffering from PTSD and SUD symptoms.
  Arms: Cognitive processing therapy
Drug: Sertraline — Sertraline for the treatment of post-traumatic stress and SU disorders
  Other Names: SSRI
  Arms: Sertraline
Other: Placebo Control — Placebo Control
  Arms: Control group

SUMMARY:
The present research was aimed at comparing the effects of Cognitive Processing Therapy (CPT) with the effects of Sertraline in treating patients who have dual diagnosis PTSD & SUD. The present study examines the extent to which CPT is effective in treating PTSD symptoms for patients with PTSD and SUD.

DETAILED DESCRIPTION:
Patients with co-occurrence PTSD & SUD disorders were grouped into 3 groups: first: Cognitive Processing Therapy (CPT) in which participants completed 12 sessions of CPT. Second: were treated by Sertraline. Third: a placebo control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with SUD

Exclusion Criteria:

* Patients diagnosed with other psychotic disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 3 Months
  A psychological parameter will be measured to check the efficacy of CPT against medication for the treatment for co-current PTSD & SUD. The groups will be examined to show if any significant reductions in PTSD and SUD symptoms was obtained over time.

CONTACTS AND LOCATIONS:
Overall Officials: Amani Elbarazi, Ph.D., Principal Investigator — The British University in Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03469128/Prot_SAP_003.pdf
  • Informed Consent Form (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03469128/ICF_004.pdf